CLINICAL TRIAL: NCT07169383
Title: Efficacy of Oral Melatonin Versus Oral Tranexamic Acid in the Management of Melasma
Brief Title: Oral Melatonin Versus Oral Tranexamic Acid in the Management of Melasma
Acronym: Melasma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Hina Malik (Other)
Responsible Party: Sponsor-Investigator, Hina Malik, Post Graduate Trainee, PAEC General Hospital, Islamabad
Organization: PAEC General Hospital, Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAECGHIslamabad
Record Dates: First submitted 2025-07-31; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Melasma (Facial Melasma)
Keywords: Management of Melasma
MeSH Terms: conditions — Melanosis | interventions — Melatonin; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Efficacy of oral melatonin and oral tranexamic acid in the management of melasma is given in patients to assess the effect of both the drugs. Two groups containing 80 participants in each. Group A is assigned oral melatonin 5mg every night for 3 months while Group B is assigned oral tranexamic acid 250mg twice daily for 3 months and then MASI score is calculated at Day One , 6 weeks and at 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Oral melatonin (Active Comparator): Group A will receive oral melatonin 5mg daily at night for 3 months after ruling out any contraindications. Melasma Area and severity index will be calculated at day one , 6 weeks and 12 weeks.
  Interventions: Drug: Melatonin tablet
- Group B - Oral tranexamic acid (Active Comparator): Group B will receive oral tranexamic acid 250mg twice daily for 3 months after ruling out any contraindications.Melasma area and severity index will than be calculated on day one , 6 weeks and 12 weeks.
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Melatonin tablet — Group A will receive oral melatonin 5mg every night for 3 months
  Arms: Group A - Oral melatonin
Drug: Tranexamic Acid (TXA) — Group B will receive oral tranexamic acid 250mg twice daily for 3 months.
  Arms: Group B - Oral tranexamic acid

SUMMARY:
This study will compare the efficacy of oral melatonin and oral tranexamic acid in treating melasma, with the aim of determining whether melatonin is more effective than tranexamic acid, as measured by MASI scores. Literature suggests melatonin may be more effective due to its antioxidant, anti-inflammatory, and anti-melanogenic properties. The findings will assess whether melatonin provides better efficacy and tolerance compared to tranexamic acid in managing this persistent condition. Efficacy will be assessed by comparing the baseline MASI scores with the scores obtained at six-week and twelve-week follow-up points based on the following cut-offs:

<25% improvement Mild response 25-50% improvement Moderate Response 51-75% improvement Good response >75% improvement Excellent Response

DETAILED DESCRIPTION:
This study will compare the efficacy of oral melatonin and oral tranexamic acid in treating melasma.Literature suggests melatonin may be more effective due to its antioxidant, anti-inflammatory, and anti-melanogenic properties.Efficacy will be assessed by comparing the baseline MASI scores with the scores obtained at six-week and twelve-week follow-up points based on the following cut-offs:

<25% improvement Mild response 25-50% improvement Moderate Response 51-75% improvement Good response >75% improvement Excellent Response It's a Randomized Control Trial conducted at PAEC General Hospital. Study period is of 6 months.Total sample size is 180 patents.The sample is divided into two groups, with 80 patients assigned to each treatment.This study hypothesizes that oral melatonin will be more effective than oral tranexamic acid in reducing the severity of melasma, as measured by changes in the Melasma Area and Severity Index.

ELIGIBILITY:
* Inclusion Criteria:

  * Adult patients aged 18-50 years diagnosed with melasma.
  * Both genders.
* Exclusion Criteria:

  * Patients with contraindications to melatonin, including pregnancy, breastfeeding, autoimmune disorders, bleeding disorders, and diabetes, or contraindications to tranexamic acid, including thromboembolic events, history of thrombosis, renal impairment, and pregnancy or breastfeeding.
  * Patients with a history of hypersensitivity to any of the medications.
  * Patients already taking treatment of melasma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Total participants are 160, 80 in Group A and 80 in Group B | 12 weeks
  Group A will receive oral melatonin 5mg HS for 12 weeks and Group B will receive oral tranexamic acid 250 mg BD for 12 weeks and then the improvement will be assessed by calculating MASI score at day 1, 6weeks and 12 weeks.MASI score less than 10 is considered mild , 11-20 is considered moderate and more than 20 is considered Severe Melasma. An improvement greater than 25% in the MASI score will be considered as the threshold for treatment efficacy.
Efficacy of Oral Melatonin VS Oral Tranexamic Acid in the management of Melasma | 12 weeks
  As per literature Melatonin may be more effective due to its Antioxidant, Anti-inflammatory and anti-melanogenic properties. The findings will assess whether Melatonin provides better efficacy and tolerance compared to Tranexamic Acid in managing Melasma.An improvement greater than 25% in the MASI score will be considered as the threshold for treatment efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- PAEC General Hospital Islamabad Pakistan, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The plan to share de-identified individual participant data (IPD) from this clinical trial, including the efficacy of oral melatonin versus oral tranexamic acid in managing melasma, with researchers who submit a methodologically sound proposal for secondary analysis. The data shared will include the primary and secondary outcome measures, participant demographics, and other relevant study data. Data will be accessible 12 months after the primary publication of the trial results, via a secure online platform, with a data use agreement. Access will be granted to researchers who provide a detailed proposal and agree to the terms of data sharing, including maintaining participant confidentiality and not attempting to re-identify participants. Requests for data access should be directed to dr.hina567@gmail.com
  This IPD sharing plan aligns with the ICMJE's expectations for data sharing and transparency in clinical trials.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2026 to janurary 2027
Access Criteria: De-identified IPD will be shared with qualified researchers who submit a proposal for secondary analysis that aligns with the trial's objectives and methodology. Proposals must outline planned analyses, including statistical methods, and will be reviewed by an independent committee for scientific merit and feasibility. A data sharing agreement must be signed, ensuring participant confidentiality and data protection. Requests can be sent to dr.hina567@gmail.com. Access will be granted for analyses that advance knowledge in melasma management, such as exploring treatment efficacy, safety, or predictors of response.

REFERENCES:
- See also: Oral Melatonin 5mg is proved to be beneficial in the management of melasma — https://pubmed.ncbi.nlm.nih.gov/38226560/
- See also: Oral Tranexamic Acid 250 mg twice a day is proved to be benefiical in the management of melasma. — https://pubmed.ncbi.nlm.nih.gov/30536592/